CLINICAL TRIAL: NCT03591185
Title: FallSensing Clinical Tool for Fall Risk Prevention in Community-dwelling Adults Aged 50 Years or Over
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anabela Correia Martins (Other)
Collaborators: Sensing Future Technologies (Other); Fraunhofer Portugal Research Center for Assistive Information and Communication Solutions (Other)
Responsible Party: Sponsor-Investigator, Anabela Correia Martins, Senior Lecturer Physiotherapy Dept., Escola Superior de Tecnologia da Saúde de Coimbra
Organization: Escola Superior de Tecnologia da Saúde de Coimbra (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1; POCI-01-0247-FEDER-003464 (Other Grant/Funding Number: Co-funded by Portugal 2020 framed under the COMPETE 2020 and European Regional Development Fund (ERDF) from EU.)
Record Dates: First submitted 2018-06-04; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Accidental Falls
Keywords: Accidental Falls; Primary prevention; Pressure platform; Inertial Sensor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise group (Experimental): Exercise group, including community-dwelling adults aged 50 years or over, will perform an initial evaluation, 24 intervention sessions with FallSensing clinical tool (2 or 3 sessions per week) and a final evaluation.
  Interventions: Other: FallSensing Clinical Tool

INTERVENTIONS:
Other: FallSensing Clinical Tool — FallSensing clinical tool will be applied to a group of community-dwelling adults aged 50 years or over, including a initial evaluation, 24 intervention sessions (2 or 3 sessions per week) and a final evaluation.
  Inicial and final evaluation consists in six functional tests (Grip Strength, Timed Up and Go, 30 seconds Sit-to-Stand, Step test, 4 Stage Balance test "modified" and 10 meters Walking Speed) and a questionnaire concerning self-efficacy for exercise.

SUMMARY:
Fall prevention programs should include strength and balance training, home hazard assessment and intervention, vision assessment and referral and also medication review with modification/withdrawal. Evidence exists that a tailored exercise program can reduce falls by as much as 54%.

Several studies recognize the benefits of the Otago Exercise Program (OEP) on physical functioning and falls reduction in older people. The program includes strength and balance exercises with a difficulty level progression by increasing weights and number of repetitions, in association with a walking plan.

FallSensing clinical tool includes a software, a pressure platform and two inertial sensors. The software includes a range of exercises based on Otago Exercise Program, including warming, balance and strength exercises. The software allows that healthcare professional prescribes a tailored exercise program according to the individual needs. During exercise performance, pressure distribution can be analysed by the healthcare professional, providing real time feedback to the individual.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 50 years or over;
* Community-dweller
* independent to be standing and walking, with or without walking aids,
* interest to participate in the study.

Exclusion Criteria:

* individuals with severe sensorial impairments (deafness or blindness)
* individuals with cognitive impairments which precludes the ability to comprehend the questionnaire, functional tests and exercises included in the protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go | Change from baseline time to perform TUG up to 12 weeks
  seconds
Self-efficacy for Exercise | Change from baseline Self-efficacy for exercise score up to 12 weeks
  Score 5 to 20 points

SECONDARY OUTCOMES:
Grip Strength | Outset and up to 12 weeks
  Kilogram-force
30 seconds Sit-to-Stand | Outset and up to 12 weeks
  number of stands
Step Test | Outset and up to 12 weeks
  number of steps
4 Stage Balance Test "Modified" | Outset and up to 12 weeks
  last position accomplished
10 meters Walking Speed | Outset and up to 12 weeks
  meters per second

CONTACTS AND LOCATIONS:
Locations (1):
- Physio Mondego, Coimbra, Portugal